CLINICAL TRIAL: NCT07051070
Title: Efficacy and Safety of Rituximab in the Treatment of Anti-Vimentin Antibody-associated Diseases
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025XW-VIMA
Record Dates: First submitted 2025-06-16; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Anti-Vimentin Antibody-associated Diseases; Meningoencephalomyelitis Associated With Vimentin IgG Autoantibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RTX treatment group (Other): This study used a drug dosage based on previous domestic and international literature as well as clinical experience from our center, set at 375mg/m2 per dose. During the course of the disease, TB lymphocyte subsets are monitored, and if the proportion of B lymphocytes is greater than or equal to 1%, a second dose will be administered.
  Interventions: Drug: RTX treatment

INTERVENTIONS:
Drug: RTX treatment — This study used a drug dosage based on previous domestic and international literature as well as clinical experience from our center, set at 375mg/m2 per dose. During the course of the disease, TB lymphocyte subsets are monitored, and if the proportion of B lymphocytes is greater than or equal to 1%, a second dose will be administered.

SUMMARY:
In 2025, a novel meningoencephalomyelitis associated with Vimentin IgG in cerebrospinal fluid (CSF) has been identified. Most patients exhibited progressive or recurrent episodes, characterized by prominent cerebellar ataxia, cranial nerve palsies, and pyramidal signs. The characteristic features included bilateral magnetic resonance imaging (MRI) lesions of the corticospinal tract, elevated CSF protein levels, and increased CSF cell counts. Despite receiving immunotherapy, these patients experienced significant disability.

This study employed a single-center, open-label, single-arm design to investigate the clinical efficacy and safety of rituximab (RTX) treatment in 40 patients with vimentin antibody (VIMA)-related diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, no gender restrictions;
2. Patients with positive CSF anti-Vimentin antibodies（VIMA）, clinically consistent with the clinical features of VIMA-related diseases reported in JAMA Neurology 2024; 3. EDSS ≥ 3.5 points or evidence of disease activity as defined by the protocol within 1 year prior to screening.

Evidence of disease activity as defined by the protocol: One of the following manifestations within 6 months of the screening period: 1. Enlargement of lesions on brain or spinal cord MRI T2 sequence; 2. △EDSS > 0; 3. At least two FS scores increase by 1 point or at least 1 FS increases by 2 points (excluding rectal/bladder and brain); 4. Symptoms lasting for more than 24 hours without fever and more than 30 days since the last episode. 4. Sign informed consent.

Exclusion Criteria:

1. Allergy to the study drug;
2. Known active infections during the screening period (excluding nail bed fungal infections or dental caries);
3. Underwent any surgical procedure within 4 weeks prior to screening, has evidence of other demyelinating diseases or progressive multifocal leukoencephalopathy (PML);
4. Positive serology for HIV or syphilis treponema or RPR during the screening period (if syphilis antibodies are negative, further serological testing for syphilis is not required);
5. Chronic hepatitis B virus or hepatitis C virus infection that meets the following criteria: • HBsAg positive; • If HBsAg negative, HbcAb positive, further HBV DNA testing (result ≥1000 IU/mL); • If HCV antibody testing is positive, further HCV RNA testing (result above the upper limit of normal range at the research site);
6. Evidence of active tuberculosis (excluding patients receiving medication for latent TB infection);
7. Received any live vaccine or attenuated live vaccine within 6 weeks prior to the medication;
8. History of malignant tumors within 5 years prior to screening, including solid tumors, hematological malignancies, and carcinoma in situ (excluding fully resected and cured basal cell carcinoma, squamous cell carcinoma, and cervical carcinoma in situ);
9. Pregnant or breastfeeding women; for women of childbearing potential, a positive serum pregnancy test at screening, or unwilling to use reliable contraception (physical barriers [patient or partner] and spermicide, contraceptive pills, patches, injections, intrauterine devices or systems), and continuing for at least 4 months after the last administration of the study drug. Men of childbearing potential unwilling to use effective contraceptive measures during the period from signing the informed consent to 6 months after the last medication;
10. Any other diseases determined by the investigator that would make the subject unsuitable for participation in this study;
11. Presence of the following clinically significant diseases:

    1. Echocardiography during the screening period shows a left ventricular ejection fraction (EF) below 50% or below the lower limit of normal values at the research center; history of chronic congestive heart failure, functional class NYHA III-IV;
    2. Any of the following events occurred within 3 months prior to signing the informed consent: myocardial infarction, acute coronary syndrome, viral myocarditis, pulmonary embolism, stroke; coronary revascularization surgery within 6 months;
    3. Electrocardiogram during the screening period indicates QTc interval >480ms (according to Fridericia's correction formula, where QTc=QT/RR^0.33), or history of severe QTc interval prolongation;
12. Laboratory test values during the screening period show the following abnormalities:

    1. Aspartate aminotransferase (AST) > 3× upper limit of normal (ULN), alanine aminotransferase (ALT) > 3× ULN, total bilirubin > 1.5× ULN (unless due to Gilbert's syndrome);
    2. Platelet count <50,000/μL (or <50 × 10^9/L), hemoglobin <9 g/dL (or <90 g/L), white blood cells <2.0 × 10^3/μL, absolute neutrophil count <1.0 × 10^3/μL;
    3. Creatinine clearance (CLcr) <60 mL/min (calculated using the Cockcroft-Gault formula: [140 - age (years)] × [weight (kg)] × (0.85, if female) / [72 × serum creatinine (mg/dL)]) or undergoing dialysis during screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Expanded Disability Status Scale (EDSS) score from baseline | baseline, week 48 after treatment.
  Change in Expanded Disability Status Scale (EDSS) score from baseline at week 48 after treatment (EDSS:Minimum Score 0, Maximum score 10, higher scores mean a worse outcome)

SECONDARY OUTCOMES:
Annualized Relapse Rate (ARR) | Week 48 after treatment
  ARR is lower, the better.
The event of confirmed disability progression (CDP) | Week 48 after treatment
  An increase of ≥1.0 points for baseline EDSS scores ≤5.5, or an increase of ≥0.5 points for baseline EDSS >5.5 is referred to as CDP.
Change in modified Rankin Scale (mRS) score from baseline | baseline, week 48 after treatment
  Change in modified Rankin Scale (mRS) score from baseline at week 48 after treatment (mRS: Minimum Score 0, Maximum score 6, higher scores mean a worse outcome )
Change in time taken to complete the Timed 25-Foot Walk (T25FW) from baseline | baseline, week 48 after treatment
  Change in time taken to complete the Timed 25-Foot Walk (T25FW) from baseline at week 48 after treatment. The time of T25FW is shorter, the better.
Change in EQ-5D-5L scores from baseline | baseline, week 48 after treatment
  Change in EQ-5D-5L scores from baseline at week 48 after treatment(EQ-5D-5L: Minimum Score 5, Maximum score 25, lower scores mean a better quality of life )
Changes in scale for the assessment and rating of ataxia (SARA) from baseline | baseline, week 48 after treatment
  Changes in scale for the assessment and rating of ataxia (SARA) from baseline at week 48 after treatment(SARA: Minimum Score 0, Maximum score 40, higher scores mean a worse outcome)
Change in Scores of International Cooperative Ataxia Rating Scale (ICARS) from baseline | baseline, week 48 after treatment
  Change in Scores of International Cooperative Ataxia Rating Scale (ICARS) from baseline at week 48 after treatment(ICARS: Minimum Score 0, Maximum Score 100, higher scores mean a worse outcome)
Number of New, and/or Enlarging T2 Hyperintense Lesions Detected by Magnetic Resonance Imaging (MRI) of brain and spinal cord | baseline, week 48 after treatment
  Number of new, and/or enlarging T2 hyperintense lesions detected by Magnetic Resonance Imaging (MRI) of brain and spinal cord at week 48 after treatment
Adverse events | through study completion, an average of 2 year
  Adverse events during use of RTX

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No